CLINICAL TRIAL: NCT05032495
Title: Patient Directed Strategies for Cardiac Arrhythmia
Brief Title: Patient Engagement Study to Evaluate the Use of Biological Therapies for Cardiac Arrhythmias
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Darryl Davis, Principal Investigator, Ottawa Heart Institute Research Corporation
Other Study IDs: 3174
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Arrythmia
Keywords: Patient engagement
MeSH Terms: conditions — Arrhythmias, Cardiac; Patient Participation | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Heart patients who experienced a cardiac arrhythmia while in hospital: Heart patients who experienced a cardiac arrhythmia while in hospital
  Interventions: Other: Surveys; Other: Focus group
- Heart patients who did not experience a cardiac arrhythmia while in hospital: Heart patients who did not experience a cardiac arrhythmia while in hospital
  Interventions: Other: Surveys; Other: Focus group
- Heart patients with an upcoming procedure that have not had a cardiac arrhythmia: Heart patients with an upcoming procedure that have not had a cardiac arrhythmia
  Interventions: Other: Surveys; Other: Focus group
- Members of the general public: Members of the general public
  Interventions: Other: Surveys; Other: Focus group

INTERVENTIONS:
Other: Surveys — Surveys to evaluate prior experience, opinions and intervention acceptability.
Other: Focus group — To answer any questions and discuss topics covered in the standard presentation.

SUMMARY:
In this patient engagement study, patients and partners will attend a presentation, group meeting and responding to the survey to help the research team gage the acceptability of using a biological therapy to prevent cardiac arrhythmia. Patient Partners will also help to clarify which outcomes are important to patients, to ensure the selected outcomes align with patient interests.

DETAILED DESCRIPTION:
There will be four study groups:

1. Heart patients who experienced a cardiac arrhythmia while in hospital,
2. Heart patients who did not experience a cardiac arrhythmia while in hospital,
3. Heart patients with an upcoming procedure that have not had a cardiac arrhythmia,
4. Members of the general public.

There will be a presentation, two surveys and a team meeting. Results will be compiled and analyzed.

ELIGIBILITY:
Inclusion criteria:

* Upcoming or previous cardiac procedure.

Exclusion Criteria:

* Inability to complete an electronic survey or participate in a small group meeting.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from in house databases after confirming patients have agreed to participate in research.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants that would accept a biological therapy for a cardiac arrhythmia as assessed using a survey | 2 years
  accept a biological therapy

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Davis, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insitute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Smith C, Lalu MM, Davis DR. Exploring Patient Viewpoints to Optimize Implementation of a Biological Therapy for Atrial Fibrillation Prevention. CJC Open. 2024 Apr 16;6(7):893-900. doi: 10.1016/j.cjco.2024.04.003. eCollection 2024 Jul. PMID 39026620